CLINICAL TRIAL: NCT06383650
Title: Use of 81 vs 325mg of ASA in Treatment of BCVI: A Feasibility RCT
Brief Title: Use of 81 vs 325mg of ASA in Treatment of BCVI
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Collaborators: Western University (Other)
Responsible Party: Principal Investigator, Kelly Vogt, Medical Director, Trauma Program, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 124532
Record Dates: First submitted 2024-03-11; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Carotid Artery Injuries; Traumatic Injury; Vertebral Artery Injury
MeSH Terms: conditions — Carotid Artery Injuries; Wounds and Injuries | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASA 81mg (Experimental): Daily study drug (x30 days)
  Interventions: Drug: Acetylsalicylic Acid
- ASA 325mg (Experimental): Daily study drug (x30 days)
  Interventions: Drug: Acetylsalicylic Acid

INTERVENTIONS:
Drug: Acetylsalicylic Acid — Patients will undergo CT imaging with the use of contrast for diagnosis of BCVI. Patients will be monitored for feasibility outcomes, as well as the development of stroke and bleeding complications.

SUMMARY:
Blunt cerebrovascular injury (BCVI), or injury to the carotid and vertebral arteries, occurs in 1-3% of blunt traumas, often as a result of injury to the head, neck, or chest. If unrecognized or untreated, BCVI can lead to stroke, which occurs in approximately 20% of untreated patients, potentially causing significant and sometimes permanent disability. Early diagnosis and treatment significantly reduce the risk of stroke.

Currently, there is wide variation across centers and trauma care providers in treatment strategies for BCVI and the most recent guidelines are unable to make specific recommendations about the optimal agent and/or dose of treatment to reduce the risk of stroke after BCVI while minimizing bleeding complications in patients with multiple traumatic injuries. Recent systematic reviews and meta-analyses evaluating the most common treatment strategies for BCVI have shown similar stroke rates with the use of anticoagulants (usually heparin) vs. antiplatelets (usually aspirin/ASA), however, treatment with antiplatelets was associated with a lower risk of bleeding complications. The optimal dose of ASA for stroke prevention while minimizing bleeding complications is unknown, and more research is required to inform future care.

This project will investigate two doses of antiplatelet therapy (81 mg daily vs. 325 mg daily aspirin) for BCVI treatment, and will look at the risk of stroke and bleeding complications with each strategy. The goal of the research is to determine whether a large-scale study looking at this question is feasible, which will ultimately help determine the best medical therapy for patients with BCVI.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Diagnosed with BCVI via CT angiography (CTA) within 72 hours of injury at a Level I Trauma Center

Exclusion Criteria:

1. ≤18 years old
2. Known Pregnancy
3. Diagnosis of BCVI made based on imaging from another hospital (non-LTH)
4. Known pre-existing carotid/vertebral artery disease
5. Stroke on presentation/before BCVI diagnosis
6. Determined to require immediate surgical or interventional management of BCVI
7. Known allergy to ASA
8. Unable to consent OR absence of a Substitute Decision Maker (SDM)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Study feasibility | 1 year
  The feasibility of the study and progression to pilot randomized controlled trial will be determined by whether it is possible to enroll ≥ 70% of eligible patients with BCVI within 90 minutes of diagnosis.

SECONDARY OUTCOMES:
Incidence of stroke | 30 days
  The secondary objective will be evaluating the effectiveness of capturing strokes in the study participants during the study period.
Incidence of Bleeding Complications | 30 days
  The secondary objective will be evaluating the effectiveness of capturing bleeding complications in the study participants during the study period.